CLINICAL TRIAL: NCT01054716
Title: Evaluation of a Noninvasive Fetal RHD Genotyping Test
Acronym: IRIS
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Sequenom Center for Molecular Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: SQNM-RHD-105
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Rhesus D Genotype
Keywords: RhD negative; RhD disease; fetal nucleic acid; fetal DNA; cell free fetal DNA; Fetal RHD genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood collected, processed to plasma and buffy coat for DNA extraction.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will collect whole blood samples from pregnant subjects who are RhD negative by serology to develop an assay for RHD determination of the fetus.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-64 years of age
* Subject is female
* Subject is pregnant
* Subject is RhD negative
* Subject is between 10 and 28 weeks gestation
* Subject provides informed consent
* Subject agrees to provide neonatal RHD and sex outcome

Exclusion Criteria:

* None

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant subjects who are RhD negative and between 10 and 28 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Fetal RHD determination from maternal whole blood | Between 10 and 28 weeks gestation

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sharp Grossmont Hospital, San Diego, California
  - West Coast OBGYN, San Diego, California
  - Women's Health Care, Inc, San Diego, California
  - Scripps Hospitals (5 San Diego locations), San Diego, California
  - Spectrum Health Research, Grand Rapids, Michigan